CLINICAL TRIAL: NCT02772237
Title: The Impact of Riboflavin on Sports-related Concussion: A Randomized Control Trial
Brief Title: The Impact of Riboflavin on Sports-related Concussion
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Collaborators: James Madison University (Other)
Responsible Party: Principal Investigator, Jeremy Kent, MD, Assistant Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18882
Record Dates: First submitted 2016-05-12; First posted 2016-05-13 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Sports-related Concussion
Keywords: concussion; sports-related concussion; mTBI; Riboflavin; Vitamin B2
MeSH Terms: conditions — Brain Concussion | interventions — Riboflavin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment group (Active Comparator): Riboflavin 400mg daily
  Interventions: Biological: Riboflavin
- Placebo group (Placebo Comparator): Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Riboflavin — Riboflavin 400mg daily
  Other Names: Vitamin B2
  Arms: Treatment group
Biological: Placebo
  Arms: Placebo group

SUMMARY:
The purpose of this study is to investigate the effectiveness of riboflavin to decrease the duration of time for a student-athlete to return to participation in sports after a sports related concussion.

ELIGIBILITY:
Inclusion Criteria:

* All UVa and JMU student-athletes over the age of 18 years old who are diagnosed with a sports related concussion

Exclusion Criteria:

* Less than 18 years old
* Greater than 24 hours have elapsed since the concussion occurred.
* The student-athlete has already participated in the study during which he/she took Riboflavin
* Non-sports related concussion not incurred while participating in the sport or training for the sport. As an example, a student-athlete who sustains a concussion as a result of a motor vehicle accident will be excluded from the study for that concussion.
* A previous concussion within the last 12 months.
* Any concussion that is complicated by a cranial bleed, skull fracture, additional severe injury (e.g. torn knee ligament) that might affect the return to normal activities above and beyond the sport-related concussion.
* If the student athlete is cognitively impaired to a level that prevents verbal communication, the consent will be deemed 'opted out' and the student-athlete will not be enrolled in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Time to return to participation in sports after a sports-related concussion | 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barbre AB, Hoane MR. Magnesium and riboflavin combination therapy following cortical contusion injury in the rat. Brain Res Bull. 2006 May 31;69(6):639-46. doi: 10.1016/j.brainresbull.2006.03.009. Epub 2006 Apr 3. PMID 16716831
- [Background] Kokiko ON, Hamm RJ. A review of pharmacological treatments used in experimental models of traumatic brain injury. Brain Inj. 2007 Mar;21(3):259-74. doi: 10.1080/02699050701209964. PMID 17453754
- [Background] Sorden SD, Lemanske RF Jr, Castleman WL. Pulmonary eosinophilia and granulomatous pulmonary arteritis induced in rats by intravenous Sephadex. Vet Pathol. 1990 Jul;27(4):217-22. doi: 10.1177/030098589002700401. PMID 1698322
- [Background] MacLennan SC, Wade FM, Forrest KM, Ratanayake PD, Fagan E, Antony J. High-dose riboflavin for migraine prophylaxis in children: a double-blind, randomized, placebo-controlled trial. J Child Neurol. 2008 Nov;23(11):1300-4. doi: 10.1177/0883073808318053. PMID 18984840
- [Background] Maizels M, Blumenfeld A, Burchette R. A combination of riboflavin, magnesium, and feverfew for migraine prophylaxis: a randomized trial. Headache. 2004 Oct;44(9):885-90. doi: 10.1111/j.1526-4610.2004.04170.x. PMID 15447697
- [Background] McCrory P, Meeuwisse W, Aubry M, Cantu B, Dvorak J, Echemendia R, Engebretsen L, Johnston K, Kutcher J, Raftery M, Sills A, Benson B, Davis G, Ellenbogen R, Guskiewicz K, Herring SA, Iverson G, Jordan B, Kissick J, McCrea M, McIntosh A, Maddocks D, Makdissi M, Purcell L, Putukian M, Schneider K, Tator C, Turner M. Consensus statement on Concussion in Sport--the 4th International Conference on Concussion in Sport held in Zurich, November 2012. J Sci Med Sport. 2013 May;16(3):178-89. doi: 10.1016/j.jsams.2013.02.009. Epub 2013 Mar 29. No abstract available. PMID 23541595
- [Background] Patterson ZR, Holahan MR. Understanding the neuroinflammatory response following concussion to develop treatment strategies. Front Cell Neurosci. 2012 Dec 12;6:58. doi: 10.3389/fncel.2012.00058. eCollection 2012. PMID 23248582
- [Background] Schoenen J, Jacquy J, Lenaerts M. Effectiveness of high-dose riboflavin in migraine prophylaxis. A randomized controlled trial. Neurology. 1998 Feb;50(2):466-70. doi: 10.1212/wnl.50.2.466. PMID 9484373
- [Background] Sundaram U. Regulation of intestinal vitamin B(2) absorption. Focus on "Riboflavin uptake by human-derived colonic epithelial NCM460 cells". Am J Physiol Cell Physiol. 2000 Feb;278(2):C268-9. doi: 10.1152/ajpcell.2000.278.2.C268. No abstract available. PMID 10666021
- [Background] Trojian TH, Jackson E. Omega-3 polyunsaturated fatty acids and concussions: treatment or not? Curr Sports Med Rep. 2011 Jul;10(4):180-5. doi: 10.1249/JSR.0b013e31822458d5. No abstract available. PMID 23531891
- [Background] Yee AJ. Effectiveness of high-dose riboflavin in migraine prophylaxis. Neurology. 1999 Jan 15;52(2):431-2. doi: 10.1212/wnl.52.2.431-a. No abstract available. PMID 9932987